CLINICAL TRIAL: NCT00401128
Title: Phase II Study of Gemcitabine Plus Irinotecan in Patients With Metastatic Renal Cell Carcinoma
Brief Title: Gemcitabine and Irinotecan in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE-CCF-6695; P30CA043703 (NIH); CASE-CCF-6695
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Kidney Cancer
Keywords: clear cell renal cell carcinoma; recurrent renal cell cancer; papillary renal cell carcinoma; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Gemcitabine; Irinotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects and how well giving gemcitabine together with irinotecan works in treating patients with metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in patients with epithelial (clear or nonclear cell) renal cell carcinoma (RCC) treated with gemcitabine hydrochloride and irinotecan hydrochloride.
* Compare the response in patients with clear cell RCC vs nonclear cell RCC treated with this regimen.
* Determine the toxicities of this regimen.

OUTLINE: This is an open-label study.

Patients receive gemcitabine hydrochloride IV over 30 minutes and irinotecan hydrochloride IV over 90 minutes on days 1 and 8. Treatment repeats every 21 days for at least 6 courses in the absence of unacceptable toxicity or disease progression.

After completion of study treatment, patients are followed every 3 months for 1 year.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed epithelial renal cell carcinoma (RCC), including either clear cell or nonclear cell RCC
* Strong clinical evidence or biopsy proof of metastases to a site or sites distant from the primary tumor
* Measurable disease
* No untreated or progressive CNS metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy > 3 months
* Absolute neutrophil count > 1,500/mm³
* Platelet count > 100,000/mm³
* Hemoglobin > 9.5 g/dL
* Creatinine ≤ 1.8 mg/dL
* Bilirubin < 1.5 mg/dL
* Calcium < 11.5 mg/dL
* ALT and AST < 3 times upper limit of normal
* No history of any of the following:

  * Serious cardiac arrhythmia or cardiac arrhythmia requiring treatment
  * Congestive heart failure
  * Angina pectoris
  * Other severe cardiovascular disease producing limitations of physical activity (i.e., New York Heart Association class III-IV heart disease)
* No other prior malignancy except for the following:

  * Basal cell or squamous cell carcinoma of the skin
  * Carcinoma in situ of the uterine cervix
  * Any malignancy treated with curative intent and in complete remission for > 3 years
* No active peptic ulcer disease, inflammatory bowel disease, or chronic diarrhea
* No local or systemic infections requiring IV antibiotics within the past 28 days
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* Recovered from prior hormonal therapy, radiotherapy, biologic therapy, or chemotherapy
* No more than 3 prior therapeutic regimens for metastatic disease
* No prior organ allograft
* More than 28 days since prior major surgery requiring general anesthesia
* More than 28 days since prior radiotherapy to control pain from skeletal lesions
* More than 28 days since prior hormonal treatment

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-05; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Overall response
Safety and efficacy

SECONDARY OUTCOMES:
Difference in response to therapy in patients with clear vs nonclear cell renal cell carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M. Bukowski, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Case Comprehensive Cancer Center, Cleveland, Ohio, United States